CLINICAL TRIAL: NCT00756665
Title: Canary Prostate Active Surveillance Study
Brief Title: Prostate Active Surveillance Study
Acronym: PASS
Status: Recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Canary Foundation (Other); Early Detection Research Network (Network)
Responsible Party: Principal Investigator, Daniel Lin, Professor, Urology, University of Washington
Other Study IDs: 33567; RG4212000 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
Keywords: prostate; cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, white cells, DNA, urine, prostate tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Prostate Active Surveillance Study (PASS) is a research study for men who have chosen active surveillance as a management plan for their prostate cancer. Active surveillance is defined as close monitoring of prostate cancer with the offer of treatment if there are changes in test results. This study seeks to discover markers that will identify cancers that are more aggressive from those tumors that grow slowly.

DETAILED DESCRIPTION:
This is a multi-center, prospective active surveillance study with selective intervention in patients with previously untreated, clinically localized prostate cancer at diagnosis. Candidates are assessed based on an extended core biopsy, serum PSA (including PSA kinetics, if available), digital rectal examination (DRE), and assessment of cancer grade and extent.

Active surveillance is defined as serial PSA measurements and prostate examination with routine prostate biopsy and therapeutic intervention considered at the time one or more of the following:

* Grade or volume progression
* Clinical progression

The objectives of the study are as follows:

Primary Objective

• To discover and confirm biomarkers that predict aggressive disease as defined by pre-specified histological, PSA, clinical criteria, or outcomes based on these variables.

Secondary Objectives

* To determine the proportion of patients on active surveillance who progress based on the above criteria.
* To determine the clinical predictors of disease progression.
* To measure the recurrence-free, disease-specific, and overall survival of men on active surveillance for clinically localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate from a prostate biopsy.
* Clinically localized prostate cancer: T1-2, NX or N0, MX or M0.
* No previous treatment for prostate cancer (including hormonal therapy, radiation therapy, surgery, or chemotherapy).
* ECOG Performance Status 0 or 1.
* Patient has elected Active Surveillance as preferred management plan for prostate cancer.
* Patient consent has been obtained according to local Institutional Review Board for acquisition of research specimens.
* Patient is accessible and compliant for follow-up.
* Prostate cancer diagnosis cannot be more than 3 years prior to baseline visit date.
* No more than two prostate biopsies including the initial biopsy in which cancer was diagnosed.
* If cancer diagnosis is more than one year before enrollment, there must be two prostate biopsies including the initial biopsy in which cancer was diagnosed and a subsequent biopsy. The subsequent biopsy may occur on the same day as the baseline visit.
* Biopsies must have at least 10 cores.

Exclusion Criteria:

* Unwillingness or inability to undergo serial prostate biopsy.
* History of other malignancies, except: adequately treated non-melanoma skin cancer or adequately treated superficial bladder cancer (Ta) or other solid tumors curatively treated with no evidence of disease for > 5 years.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Urology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2008-07; Primary Completion 2029-09 (Estimated); Study Completion 2032-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W. Lin, MD, Principal Investigator — University of Washington; James D. Brooks, MD, Principal Investigator — Stanford University; Martin E. Gleave, MD, Principal Investigator — University of British Columbia; Michael Liss, MD, Principal Investigator — University of Texas Health Science Center San Antonio; Peter R. Carroll, MD, MPH, Principal Investigator — University of California, San Francisco; Robert W. Given, MD, Principal Investigator — Eastern Virginia Medical School; Andrew A Wagner, MD, Principal Investigator — Beth Israel Deaconess Medical Center/Harvard Medical School; Todd M. Morgan, MD, Principal Investigator — University of Michigan; Lisa F Newcomb, PhD, Study Director — Fred Hutchinson Cancer Research Center/University of Washington; Martin G. Sanda, MD, Principal Investigator — Emory University; Matthew R. Cooperberg, MD, MPH, Principal Investigator — Veterans Affairs San Francisco Health Care System; Atreya Dash, MD, Principal Investigator — Veterans Affairs Puget Sound Health Care System
Locations (11):
- United States (10):
  - Veterans Affairs San Francisco Health Care System, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Emory University, Atlanta, Georgia
  - Beth Israel Deaconess Medical Center/Harvard Medical School, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Texas Health Science Center, San Antonio, San Antonio, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Veterans Affairs Puget Sound Health Care System, Seattle, Washington
  - University of Washington, Seattle, Washington
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Warlick CA, Allaf ME, Carter HB. Expectant treatment with curative intent in the prostate-specific antigen era: triggers for definitive therapy. Urol Oncol. 2006 Jan-Feb;24(1):51-7. doi: 10.1016/j.urolonc.2005.07.004. PMID 16414495
- [Background] Carter HB, Walsh PC, Landis P, Epstein JI. Expectant management of nonpalpable prostate cancer with curative intent: preliminary results. J Urol. 2002 Mar;167(3):1231-4. PMID 11832703
- [Background] Hardie C, Parker C, Norman A, Eeles R, Horwich A, Huddart R, Dearnaley D. Early outcomes of active surveillance for localized prostate cancer. BJU Int. 2005 May;95(7):956-60. doi: 10.1111/j.1464-410X.2005.05446.x. PMID 15839912
- [Background] Klotz L. Active surveillance with selective delayed intervention for favorable risk prostate cancer. Urol Oncol. 2006 Jan-Feb;24(1):46-50. doi: 10.1016/j.urolonc.2005.07.002. PMID 16414494
- [Background] Meng MV, Elkin EP, Harlan SR, Mehta SS, Lubeck DP, Carroll PR. Predictors of treatment after initial surveillance in men with prostate cancer: results from CaPSURE. J Urol. 2003 Dec;170(6 Pt 1):2279-83. doi: 10.1097/01.ju.0000094190.46523.b2. PMID 14634396
- [Background] Patel MI, DeConcini DT, Lopez-Corona E, Ohori M, Wheeler T, Scardino PT. An analysis of men with clinically localized prostate cancer who deferred definitive therapy. J Urol. 2004 Apr;171(4):1520-4. doi: 10.1097/01.ju.0000118224.54949.78. PMID 15017211
- [Background] Roemeling S, Roobol MJ, de Vries SH, Wolters T, Gosselaar C, van Leenders GJ, Schroder FH. Active surveillance for prostate cancers detected in three subsequent rounds of a screening trial: characteristics, PSA doubling times, and outcome. Eur Urol. 2007 May;51(5):1244-50; discussion 1251. doi: 10.1016/j.eururo.2006.11.053. Epub 2006 Dec 5. PMID 17161520
- [Background] Kattan MW, Eastham JA, Wheeler TM, Maru N, Scardino PT, Erbersdobler A, Graefen M, Huland H, Koh H, Shariat S, Slawin KM, Ohori M. Counseling men with prostate cancer: a nomogram for predicting the presence of small, moderately differentiated, confined tumors. J Urol. 2003 Nov;170(5):1792-7. doi: 10.1097/01.ju.0000091806.70171.41. PMID 14532778
- [Background] Steyerberg EW, Roobol MJ, Kattan MW, van der Kwast TH, de Koning HJ, Schroder FH. Prediction of indolent prostate cancer: validation and updating of a prognostic nomogram. J Urol. 2007 Jan;177(1):107-12; discussion 112. doi: 10.1016/j.juro.2006.08.068. PMID 17162015